CLINICAL TRIAL: NCT06879002
Title: To Compare IVF/ICSI Cycle Outcomes of Post Ovulation Ovarian Stimulation Protocol With Elonva Without GnRH Antagonist to Follicular Phase Fixed Day 5 Antagonist Protocol
Brief Title: Comparing IVF/ICSI Cycle Outcomes of Post Ovulation Ovarian Stimulation Protocol With Elonva Without GnRH Antagonist to Follicular Phase Day 2 Stimulation Fixed Day 5 Antagonist Protocol
Status: Not yet recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Maryam Farid Mojtahedi, Specialist IVF, ART Fertility Clinics LLC
Other Study IDs: 2409-ABU-015-MF
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-06

CONDITIONS: Stimulation in the Ovary; IVF Outcome
Keywords: progesterone; premature ovulation; ovarian stimulation; luteal stimulation
MeSH Terms: interventions — Ovulation Induction; Menstruation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: - Follicular phase start of ovarian stimulation with Elonva: Patients considered for ovarian stimulation for IVF/ICSI will be informed and a CF will be given on the day of planning for IVF. In group one, the ovarian stimulation protocol would follow a fixed GnRH antagonist protocol with recombinant FSH, Corifolitropin alfa (Elova150 mcg) starting on day 2 of the menstrual cycle.
  Group A: Day 2-3 of cycle: Estradiol, Progesterone, Luteinizing Hormone, Follicle stimulating hormone During stimulation: on day 8 of stimulation: Estradiol, Progesterone, Luteinizing Hormone, Follicle stimulating hormone on trigger day: Estradiol, Progesterone, Luteinizing Hormone, Follicle stimulating hormone
  Final oocyte maturation will be administered when 3 follicles reach 17mm or more. Oocyte retrieval will be performed 36 hours after human chorionic gonadotropin (hCG5000 or 10000IU, choriomon, IBSA) plus GnRH-a (0.2 or 0.3 mg Gonapeptyl, Ferring) administration under transvaginal ultrasound guidance.
  Interventions: Other: Ovarian stimulation with menstruation or after ovulation
- Group B: One day after the Positive LH kit test at home: E2 P4 LH FSH,BHCG: . In group two, Elona 150mcg is being administered after ovulation confirmation with home LH kits starting to be used around usual ovulation days, and be confirmed in clinic with LH rise, E2 drop and blood P4 more than 1ng/dl one day after LH kit is positive. The probability of spontaneous pregnancy will be ruled out by betaHCG test. In case a spontaneous pregnancy has been confirmed,we will not start the treatment . Furthermore, in case of sustained progesterone rise,repeated hCG tests will be performed throughout the stimulation cycle to monitor whether there is an early pregnancy or not. If so,the treatment will be cancelled/stopped to prevent the potential risks of stimulation medications during an early pregnancy.From stimulation Day 8 onwards, hormonal stimulation will continue with daily dose. The maximum injection dose for continuing treatment after the first 7 days will be 200 IU. (10) Final oocyte maturation will be administered when 3 follicles reach 17mm or more.
  Interventions: Other: Ovarian stimulation with menstruation or after ovulation

INTERVENTIONS:
Other: Ovarian stimulation with menstruation or after ovulation — Ovarian stimulation with menstruation or after ovulation

SUMMARY:
There are several approaches to the timing of antagonist administration in IVF/ICSI cycles. The primary goal is indeed to prevent premature ovulation, which could jeopardize the success of the cycle There is an emerging concept that suggests that the progesterone produced by the corpus luteum (formed after ovulation) might be sufficient to prevent further ovulation, obviating the need for antagonist or exogenous progesterone administration. This hypothesis relies on the natural regulatory mechanisms of the menstrual cycle to maintain a progesterone-dominated environment post-ovulation. We hypothesized that this approach would minimize treatment costs /burden without having an impact on the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 38 years old.
* Normal Menstrual cycle of 25-35 days.
* Body Weight 60to90 kg
* AMH>1.3 - <3 ng/m (Ferraretti and Gianaroli, 2014; Calzada et al., 2019) an antral follicle count (AFC) of >5 on menstrual cycle days 2-3,

Exclusion Criteria:

* History of premature ovulation
* Azoospermia
* PCOS
* Endometriosis AFS ¾
* Endometrioma
* Known chromosomal abnormalities

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — - Expected normal responder patients who undergo IVF/ICSI+PGT-A at ART Fertility Clinics Dubai & Abu Dhabi &Alain who are willing to participate in the study after signing the Consent Form.
Study Population: Expected normal responder patients who undergo IVF/ICSI+PGT-A at ART Fertility Clinics Dubai & Abu Dhabi are willing to participate in the study.
Sampling Method: Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Oocyte maturity, Fertilization rate, Blastulation rate, quality Euploidy rate, Premature ovulation rate, Number of injections used and costs | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Study Director — ART Fertility Clinics LLC
Locations (2):
- United Arab Emirates (2):
  - ART Fertility Clinics LLC, Abu Dhabi
  - ART Fertility Clinics LLC - Dubai, Dubai

IPD SHARING:
Plan to Share IPD: Undecided
upon request

REFERENCES:
- [Background] Ata B, Kalafat E. Progestin-primed ovarian stimulation: for whom, when and how? Reprod Biomed Online. 2024 Feb;48(2):103639. doi: 10.1016/j.rbmo.2023.103639. Epub 2023 Oct 22. PMID 38159467
- [Background] Giles J, Cruz F, Garcia-Velasco JA. Progestin-primed ovarian stimulation. Curr Opin Obstet Gynecol. 2024 Jun 1;36(3):165-172. doi: 10.1097/GCO.0000000000000941. Epub 2024 Jan 30. PMID 38295019
- [Background] Glujovsky D, Pesce R, Miguens M, Sueldo CE, Lattes K, Ciapponi A. How effective are the non-conventional ovarian stimulation protocols in ART? A systematic review and meta-analysis. J Assist Reprod Genet. 2020 Dec;37(12):2913-2928. doi: 10.1007/s10815-020-01966-5. Epub 2020 Nov 21. PMID 33219862
- [Background] Kolibianakis EM, Venetis CA, Kalogeropoulou L, Papanikolaou E, Tarlatzis BC. Fixed versus flexible gonadotropin-releasing hormone antagonist administration in in vitro fertilization: a randomized controlled trial. Fertil Steril. 2011 Feb;95(2):558-62. doi: 10.1016/j.fertnstert.2010.05.052. Epub 2010 Jul 16. PMID 20637457